CLINICAL TRIAL: NCT06642753
Title: Buccal Plate Augmentation Using Sticky Bone Versus Usage of Sticky Bone as a Jumping Gap Filling Material With Simultaneous Immediate Implant Placement in the Maxillary Esthetic Zone :A Randomized Controlled Clinical Trial
Brief Title: Buccal Plate Augmentation Using Sticky Bone With Simultaneous Immediate Implant Placement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yara Khaled Mahmoud Khalefa Ghaith, Principal Investigator yara khaled Master Degree student, Periodontology department, Faculty of Dentistry, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PER.6-3-1
Record Dates: First submitted 2024-08-05; First posted 2024-10-15 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-09

CONDITIONS: Immediate Implant
Keywords: buccal plate preservation; sticky bone; PRF

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- immediate implant with buccal plate augmentation using sticky bone (Experimental): atraumatic extraction.
  * The socket will be well irrigated with saline and debrided with a bone curette.
  * placement of the implant.
  * Venous blood will be withdrawn and transferred into sterile tubes which will be devoid of anticoagulants. I- PRF preparation will be done using the protocol developed by Mourãoet al.
  * sticky bone will be ready to be grafted.
  * Sticky bone will be inserted into the pouch by a mean of a small periosteal elevator. Additional graft material will be added and compressed until adequate filling of the pouch is achieved without overstretching the soft tissues.
  * the healing abutment will be screwed into the implant body .
  Interventions: Biological: immediate implant with buccal plate augmentation using sticky bone
- immediate implant with sticky bone as a filling material in the jumping gap (Active Comparator): * atraumatic extraction.
  * The socket will be well irrigated with saline and debrided with a bone curette.
  * placement of the implant.
  * Venous blood will be withdrawn and transferred into sterile tubes which will be devoid of anticoagulants. I- PRF preparation will be done using the protocol developed by Mourãoet al.
  * sticky bone will be ready to be grafted.
  * The sticky bone graft will be condensed and adapted into the jumping gap as well as over the implants. Further, it will be covered with PRF membrane.
  * the healing abutment will be screwed into the implant body
  Interventions: Biological: immediate implant with sticky bone as a filling material in the jumping gap

INTERVENTIONS:
Biological: immediate implant with buccal plate augmentation using sticky bone — * Venous blood will be withdrawn and transferred into sterile tubes which will be devoid of anticoagulants. I- PRF preparation will be done using the protocol developed by Mourãoet al.
  * Plastic PET tubes to create Liquid-PRF, while glass tubes will be used to obtain Solid-PRF.
  * Blood will be centrifuged at a speed of 3000 rpm for 10 minutes to obtain autologous PRF plug.
  * Blood will be centrifuged at a speed of 700 rpm for 3 minutes. An orange- colored fluid will be formed as the upper layer in the test tubes i.e., I- PRF. Approximately 1 ml of I-PRF will be collected in a syringe.
  * Solid-PRF + Liquid-PRF mixed DBBM: Solid-PRF membranes will be mixed thoroughly with 0.25 g of DBBM particles. Then 1 mL Liquid PRF from the buffy coat layers will be added drop by drop to the DBBM.
  * Following polymerization by 15-20 minutes, sticky bone will be ready to be grafted in the pouch .
  Arms: immediate implant with buccal plate augmentation using sticky bone
Biological: immediate implant with sticky bone as a filling material in the jumping gap — Venous blood will be withdrawn and transferred into sterile tubes which will be devoid of anticoagulants. I- PRF preparation will be done using the protocol developed by Mourãoet al.
  * Plastic PET tubes to create Liquid-PRF, while glass tubes will be used to obtain Solid-PRF.
  * Blood will be centrifuged at a speed of 3000 rpm for 10 minutes to obtain autologous PRF plug.
  * Blood will be centrifuged at a speed of 700 rpm for 3 minutes. An orange- colored fluid will be formed as the upper layer in the test tubes i.e., I- PRF. Approximately 1 ml of I-PRF will be collected in a syringe.
  * Solid-PRF + Liquid-PRF mixed DBBM: Solid-PRF membranes will be mixed thoroughly with 0.25 g of DBBM particles. Then 1 mL Liquid PRF from the buffy coat layers will be added drop by drop to the DBBM.
  * Following polymerization by 15-20 minutes, sticky bone will be ready to be grafted in the jumping gap.
  Arms: immediate implant with sticky bone as a filling material in the jumping gap

SUMMARY:
the aim of this study is to clinically assess pink esthetic score following Buccal Plate Augmentation using Sticky Bone versus usage of Sticky Bone as a jumping gap filling material with simultaneous immediate implant placement in the maxillary esthetic zone

DETAILED DESCRIPTION:
All patients will undergo pre-operative clinical examination: Patient's data will be collected; name, gender and age, medical and dental histories will be taken. Also, all patients will undergo standardized periapical radiograph to detect any pathosis and a pre-operative Cone beam computed tomography (CBCT) scans will be taken to evaluate the tooth root configuration and to confirm the presence of intact buccal wall, Vital structures related to the tooth, Vertical and horizontal dimensions of the alveolar bone and Bone density.

Patient preparation for surgical procedure:

After extra oral disinfection of the surgical site ,the patients will be asked to rinse their mouths with Chlorohexidine HCL 1.25% mouthwash (Orovex mouthwash, Macro group, Egypt) immediately preoperatively. Local infiltration anesthesia [Articaine 4% 1:100,000 epinephrine] (Artinibsa 40mg/0.1 mg/Ml ˗ epinephrine 1:100000, Spain) will be used for all procedures.

Control group:

* The surgical procedure will be performed in sterile surgical field. Under local anesthesia, sharp dissection of the supracrestal fibers will be done with no.15 c scalpel blade. With the purpose of preserving the buccal and palatal bone walls, periotomes, elevators and maxillary root forceps will be used to facilitate atraumatic extraction.
* The socket will be well irrigated with saline and debrided with a bone curette. An intact buccal bone plate should be found after extraction of the tooth.
* Bony sockets will be prepared through sequential drilling for the placement of the implant.
* Achieving primary stability after implant placement will be followed by placement of cover screw.
* Venous blood will be withdrawn under aseptic conditions by veni puncture of the antecubital vein and transferred into sterile tubes which will be devoid of anticoagulants. I- PRF preparation will be done using the protocol developed by Mourãoet al.
* Plastic PET tubes to create Liquid-PRF, while glass tubes will be used to obtain Solid-PRF.
* Blood will be centrifuged at a speed of 3000 rpm for 10 minutes to obtain autologous PRF plug.
* Blood will be centrifuged at a speed of 700 rpm for 3 minutes. An orange- colored fluid will be formed as the upper layer in the test tubes i.e., I- PRF. Approximately 1 ml of I-PRF will be collected in a syringe.
* Solid-PRF + Liquid-PRF mixed DBBM: Solid-PRF membranes will be cut into small PRF fragments sized between 1-2 mm and mixed thoroughly with 0.25 g of DBBM particles. Then 1 mL Liquid PRF from the buffy coat layers will be added drop by drop to the DBBM.
* Following polymerization by 15-20 minutes, sticky bone will be ready to be grafted.
* The sticky bone graft will be condensed and adapted into the jumping gap as well as over the implants. Further, it will be covered with PRF membrane.
* the healing abutment will be screwed into the implant body .

Intervention group:

* A thin periosteal elevator will be used to reflect the soft tissue buccal to the bony buccal plate on the mid-facial aspect of the socket in a full-thickness manner, following a corono-apical direction, thereby creating a 'surgical pouch.
* The dissection will be advanced beyond the mucogingival line to approximately two-thirds the depth of the socket, and the 'pouch' will be expanded in the mesio-distal direction to stretch the soft tissues away from the underlying bony plate.
* Sticky bone will be inserted into the pouch by a mean of a small periosteal elevator. Additional graft material will be added and compressed until adequate filling of the pouch is achieved without overstretching the soft tissues.
* the healing abutment will be screwed into the implant body .

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older.
* Presence of a non-restorable maxillary tooth in the esthetic zone including maxillary anteriors and premolars indicated for extraction.
* An intact buccal plate of bone after extraction.
* Full-mouth plaque and bleeding score not exceeding 20%.
* Patients showing motivation to comply with post-operative care instructions and follow- up appointments.

Exclusion Criteria:

* Periapical infection involving the tooth to be extracted.
* Periodontal disease
* Systemic health conditions that contraindicate or affect healing of implant surgery (Diabetes Mellitus, Leukemia)
* Pregnant and nursing females.
* Smokers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
pink esthetic score | 3 and 6 months postoperative
  This pink esthetic score (PES) evaluates the esthetic outcome of soft tissue around implant-supported single crowns in the anterior zone by awarding seven points for the mesial and distal papilla, soft-tissue level, soft-tissue contour, soft-tissue color, soft-tissue texture, and alveolar process deficiency .With the exception of papilla formation, the evaluation is performed visually by comparing reference teeth (i.e., with the contralateral tooth in the incisor zone and adjacent tooth in the premolar zone). For the mesial and distal papilla, the categories are complete, incomplete, and absent. For each criterion it is possible to award a score between two points (for a very good outcome) and no points (for a poor outcome). The maximum score that can be achieved is 14 points indicating an outcome that reflects complete conformity between the soft tissue of the tooth being assessed and that of the reference tooth.

SECONDARY OUTCOMES:
crestal bone level | baseline and 6 months post operative
  using Cone beam computed tomography (CBCT) machine with superimposition technique.
Thickness of labial plate of bone | baseline and 6 months postoperatively
  Using CBCT machine . Using the axial view, one reference line will be drawn from the apex of the implant to its platform (long axis); another line, perpendicular to the one at the long axis, will be drawn at the apex of the implant. Parallel to this, two lines will be drawn, one at 1 mm from the implant collar (R1) and another 5 mm apical to it (R2) measuring the thickness of the bone (at the buccal plate) to the nearest 0.1 mm.
Soft tissue profile /contour | baseline, 3 and 6 months postoperatively.
  Scanning of diagnostic casts by optical scanner.
patient satisfaction | immediately after implant placement , 3 and 6 months postoperative
  VAS (Visual analogue scales ) based questionnaire. for pain: The most common VAS consists of a 10-cm horizontal or vertical line with the two endpoints labeled "no pain" and "worst pain ever" (or similar verbal descriptors). The patient is required to place a mark on the 10-cm line at a point that corresponds to the level of pain intensity they presently feel. The distance in centimeters from the low end of the VAS to the patient's mark is used as a numerical index of the severity of pain.
  for swelling:
  1. no swelling.
  2. mild intraoral swelling
  3. moderate intraoral swelling
  4. severe extraoral swelling

CONTACTS AND LOCATIONS:
Overall Officials: Enji ahmed, professor, Study Director — Cairo University; shaimaa Nasr, Ass. Prof, Study Chair — Cairo University; Yara Kh Ghaith, Bachelor, Principal Investigator — Cairo University; samah bahaa, Lecturer, Study Chair — Cairo University
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Egypt

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2024-04-15): https://cdn.clinicaltrials.gov/large-docs/53/NCT06642753/Prot_ICF_001.pdf